CLINICAL TRIAL: NCT04092010
Title: Improving Preschool Outcomes by Addressing Maternal Depression in Head Start
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022003398; 1R01HD092456-01A1 (NIH)
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Maternal Depression
Keywords: Stepped care intervention; Problem solving education; Engagement session; Head Start; Preschool children

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped-care intervention (SCI) group (Experimental): In the SCI group, mothers with low baseline depressive symptoms are offered the problem-solving education (PSE) prevention intervention, and mothers with greater depressive symptoms are offered Engagement Sessions.
  Interventions: Behavioral: Problem-solving education (PSE); Behavioral: Engagement sessions
- Usual care control group (Active Comparator): Families in the control group will receive usual Head Start services.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Problem-solving education (PSE) — PSE will be offered to mothers with low baseline depressive symptoms (the first, preventive step of the SCI). PSE participants will have their symptoms assessed at each session and will convert to Engagement Sessions if they meet pre-specified 'step up' criteria.
  Arms: Stepped-care intervention (SCI) group
Behavioral: Engagement sessions — Engagement sessions will be offered to mothers with greater depressive symptoms to link them to formal mental health services (the second, referral step of the SCI)
  Arms: Stepped-care intervention (SCI) group
Behavioral: Usual care — Normal services provided children and their mothers in Head Start
  Arms: Usual care control group

SUMMARY:
Within a research network of Head Start centers in Massachusetts, an efficacy trial of a stepped-care intervention (SCI) to address maternal depression, using intervention components that both prevent depression and help those in major depressive episode (MDE) engage with care, will be conducted. Both the prevention and engagement components of the model have strong, supportive randomized trial evidence for both their efficacy and safety; but they have yet to be synthesized and tested within a coordinated intervention, applicable to a broad population base. Stepped-care interventions are commonly used in mental health service projects, in which the intensity or type of service is calibrated to the severity of illness.

DETAILED DESCRIPTION:
This research study is a community-based efficacy trial (n=388) of a stepped-care model intervention to strengthen the capacity of Head Start to address parental depression and related adversities. Head Start mothers with symptoms of depressed mood or anhedonia, and their Head Start children, are enrolled across 12 Head Start centers.

The research study aims to improve developmental outcomes for Head Start children by delivering stepped care intervention that incorporates depression prevention and linkage to formal mental health care to mothers. Mothers with low baseline depressive symptoms are offered a problem-solving intervention while mothers with greater symptoms are offered engagement sessions to link them to formal mental health services. At each problem-solving session participant's symptoms are assessed and if the symptoms meet pre-specified 'step-up' criteria, they are converted to Engagement sessions.

Over 12 months, the intervention's effect will be assessed on a series of outcome measures for mothers; mechanisms by which maternal depression is theorized to impact young children; and child outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Mother of a 0 to 5-year-old Head Start child
* Mother speaks English or Spanish

Exclusion Criteria:

* Mother with suicidal ideation
* Mother with cognitive limitation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in incident rates of moderate to severe maternal depressive symptoms based on the QIDS | Baseline, 2, 4, 6, 8, 10, 12 months follow-up
  The Quick Inventory of Depressive Symptoms (QIDS) will be used to assess the incidence of moderate to severe depressive symptom episodes, as defined by a QIDS score ≥ 11. The QIDS is a 16 item self-administered instrument with potential responses for each item of 0 to 3. Higher scores are associated with greater depressive symptoms.
Change in the mean maternal depressive symptoms based on the QIDS | Baseline, 2, 4, 6, 8, 10, 12 months follow-up
  The Quick Inventory of Depressive Symptoms will be used to assess depressive symptoms. The QIDS is a 16 item self-administered instrument with potential responses for each item of 0 to 3. Higher scores are associated with greater depressive symptoms. The mean QIDS scores will be calculated for the baseline and each follow up period.

SECONDARY OUTCOMES:
Rate of participants engaged with care based on 1 or more psycho/pharmacotherapy visits or psychiatric medication prescription | Baseline, 2, 4, 6, 8, 10, 12 months follow-up
  The investigators have adapted the services section of the Collaborative Psychiatric Epidemiology Surveys, operationalized into engagement with care. This will be defined as ≥ 1 visit for psychotherapy or pharmacotherapy with a behavioral health specialist (social worker, psychologist, psychiatrist, psychiatric nurse); or a prescription for psychiatric medication from any medical practitioner.
Rate of participants retained in care based on 4 or more psycho/pharmacotherapy visits or psychiatric medication prescription | 2, 4, 6, 8, 10, 12 months
  The investigators have adapted the services section of the Collaborative Psychiatric Epidemiology Surveys, operationalized into retention in care. This will be defined as ≥ 4 visit for psychotherapy or pharmacotherapy with a behavioral health specialist (social worker, psychologist, psychiatrist, psychiatric nurse); or a prescription for psychiatric medication from any medical practitioner.
Rate of participants who received evidence-based care defined by psychotherapy or antidepressant medication prescription | 2, 4, 6, 8, 10, 12 months
  The investigators have adapted the services section of the Collaborative Psychiatric Epidemiology Surveys, operationalized into evidence-based care reflecting either psychotherapy or antidepressant medication.
Rate of participants who received primary-care based services | 2, 4, 6, 8, 10, 12 months
  The investigators have adapted the services section of the Collaborative Psychiatric Epidemiology Surveys, operationalized into primary care-based services.
Burden of illness for depression | baseline; 6, 12 months
  The Individual Burden of Illness Index for Depression (IBI-D) is a valid and reliable quality of life (QoL) scale, calculated as a composite of the QIDS, the QoL Enjoyment and Satisfaction Questionnaire, and the Work and Social Adjustment Scale
Child absenteeism from Head Start | baseline; 6, 12 months
  Head Start centers will furnish us with monthly absentee rates for all families that provide explicit permission. These will be analyzed as count data against day of eligible attendance.
Caregiver-Teacher Report Form | baseline; 6, 12 months
  This valid and reliable scale will be filled out by Head Start teachers. It measures emotional reactivity, anxiety/depression, somatic complaints, emotional withdrawal, attention problems, and aggressive behavior.
Social Skills Improvement System - Rating Scales | baseline; 6, 12 months
  This valid and reliable scale will be filled out by Head Start teachers. It assesses social skills and problem behaviors for children at risk of interpersonal difficulties.
Bracken School Readiness Assessment | baseline; 6, 12 months
  This scale assesses 85 foundational concepts, including colors, letters, numbers, size/ comparison, and shapes. Assess effect of intervention on child cognitive functioning and school readiness.
Perceived Stress | baseline, 4, 8, 12 months
  Assess with The Perceived Stress Scale, domains of which include unpredictability, lack of control, burden overload, and stressful circumstances.
Behavioral Activation for Depression | baseline, 4, 8, 12 months
  Assess with The Behavioral Activation for Depression Scale (BADS) includes four affective and functional dimensions: activation, avoidance/rumination, work/school impairment, and social impairment.
Coping Strategies | baseline, 4, 8, 12 months
  Assess with The Brief COPE (Coping Orientation to Problems) which measures 14 different adaptive and problematic coping styles. Will also use problem-focused and avoidant subscales.
Parent-Child Interaction | baseline, 6, 12 months
  Assess with The Dyadic Parent-Child Interaction Coding System (4th Edition).
Family Conflict | Baseline, 6, 12 months
  Assess with The 80-item Conflicts and Problem-Solving Scale. Likert scales rate aspects of family conflict known to affect children: 1) number of major and minor conflicts in the past year; 2) family disagreement in 21 areas; 3) frequency of 13 conflict resolution strategies; 4) frequency of 44 conflict tactics.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Feinberg, ScD CPNP, Principal Investigator — Brown University; Michael Silverstein, MD, Principal Investigator — Brown University; Amy Yule, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data that underlie the results reported for all primary and secondary outcome measures will be made available (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 6 months after study completion and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for the purposes of reviewing proposals to gain access to these data. Requestors will need to provide a methodologically sound proposal, sign a data sharing agreement, and agree to the terms of data receipt.